CLINICAL TRIAL: NCT01845597
Title: Survivorship and Outcomes of Robotically Assisted Medial UKA
Brief Title: Survivorship and Outcomes of Robot Assisted Medial Partial Knee Replacement
Status: Completed | Type: Observational
Sponsor: Northwest Surgical Specialists, Vancouver (Other)
Collaborators: Stryker Instruments (Industry)
Responsible Party: Sponsor
Other Study IDs: MAKO-03; 2016-006 (Other: Stryker)
Record Dates: First submitted 2013-04-29; First posted 2013-05-03 (Estimated); Results first posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2022-08

CONDITIONS: Unicompartmental Knee Arthroplasty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MAKOplasty® medial UKA: Patients knees that have received a MAKOplasty® robotically guided unicompartmental knee arthroplasty (UKA) and received a medial MCK onlay implant.
  Interventions: Procedure: MAKOplasty® medial UKA

INTERVENTIONS:
Procedure: MAKOplasty® medial UKA — A robot guided medial Unicompartmental knee arthroplasty (UKA) is a procedure to replace only the medial tibiofemoral compartment of the knee.
  Other Names: Medial Partial Knee Replacement; Medial Unilateral Knee Arthroplasty; Robot Assisted Partial Knee Replacement

SUMMARY:
The purpose of this study is to determine the survivorship rate of robotic assisted medial partial knee replacement at a two, five, and ten years.

DETAILED DESCRIPTION:
The purpose of this study is to determine the survivorship rate of robotically guided MultiCompartmental Knee system (MCK) medial onlay Unicompartmental Knee Arthroplasty (UKA) implants at a two, five, and ten year follow up.

ELIGIBILITY:
Inclusion Criteria:

* over 21 years of age
* underwent primary robotically guided UKA and received a medial MCK onlay implant by the investigating surgeon
* at least 24 months post-operative

Exclusion Criteria:

* Patients will be excluded from participation in the study if they are cognitively unable to answer study questions

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent a MAKOplasty procedure by the investigating surgeon and received a medial MCK onlay implant.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2013-04; Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Borus, MD, Principal Investigator — Rebound Orthopedics and Neurosurgery
Locations (1):
- Rebound Orthopedics and Neurosurgery, Vancouver, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 179 subjects who received a robotically guided medial unicompartmental knee arthroplasty (UKA) by the investigating surgeon and were at least 2 years post-operation as of December 30, 2011. Of the 179 subjects contacted by post card and/or a phone call 145 agreed to participate in the study.
Groups:
- Robot Assisted Medial Partial Knee Replacement: Patients knees that have received a robotically guided unicompartmental knee arthroplasty (UKA) and received a medial MCK onlay implant.
  MAKOplasty® medial UKA: A robot guided medial Unicompartmental knee arthroplasty (UKA) is a procedure to replace only the medial tibiofemoral compartment of the knee.
Period: Overall Study
Arm/Group | Robot Assisted Medial Partial Knee Replacement
Started | 145
5 Year Survivorship | 134
Completed | 115
Not Completed | 30
Not completed — Death | 8
Not completed — Lost to Follow-up | 22

BASELINE CHARACTERISTICS:
Groups:
- Robot Assisted Medial Partial Knee Replacement: Patients knees that have received a MAKOplasty® robotically guided unicompartmental knee arthroplasty (UKA) and received a medial MCK onlay implant.
  MAKOplasty® medial UKA: A robot guided medial Unicompartmental knee arthroplasty (UKA) is a procedure to replace only the medial tibiofemoral compartment of the knee.
Arm/Group | Robot Assisted Medial Partial Knee Replacement
Number analyzed (Participants) | 145
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 74
  >=65 years | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.98 (8.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 80
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 145

OUTCOME MEASURES:

1. Primary Outcome: 10 Year Survivorship of Components
Description: Survivorship of components is defined as knee implant device(s) remaining in patient.
Time Frame: 10 years after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | MAKOplasty® Medial UKA
Number analyzed (Participants) | 115
Participants | 110

2. Secondary Outcome: 5 Year Survivorship of Components
Description: Survivorship of components is defined as knee implant device(s) remaining in patient.
Time Frame: 5 years after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | MAKOplasty® Medial UKA
Number analyzed (Participants) | 134
Participants | 132

3. Secondary Outcome: 2 Year Survivorship of Components
Description: Survivorship of components is defined as knee implant device(s) remaining in patient.
Time Frame: 2 years after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | MAKOplasty® Medial UKA
Number analyzed (Participants) | 145
Participants | 144

ADVERSE EVENTS:
Time Frame: 2, 5 and 10 years post surgery.
Description: The only adverse event collected was death of subject from all causes at 2, 5 and 10 years post surgery.
Arm/Group | MAKOplasty® Medial UKA
All-Cause Mortality (participants affected / at risk) | 8/145
Serious Adverse Events (participants affected / at risk) | 0/145
Other Adverse Events (participants affected / at risk) | 0/145

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2013-03-14): https://cdn.clinicaltrials.gov/large-docs/97/NCT01845597/Prot_000.pdf